CLINICAL TRIAL: NCT03880526
Title: Rural Survivorship naVigation Program (RSVP): Building Community Capacity for Cancer Control
Brief Title: Rural Survivorship Navigation Program
Acronym: RSVP
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00056939; WFBCCC 04219 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH); NCI-2019-01751 (Other: National Cancer Institute)
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: Cancer prevention control; Cancer navigation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Semi-Structured Interview: Participants will choose to participant in an individual in-depth interview to be conducted by investigators to gain information about the participant's background, cancer status and treatment.
- Focus Groups: Participants may choose to participate in one of three focus groups of no more than 10 participants in each group to to gain information about the participant's background, cancer status and treatment.

SUMMARY:
The purpose of this proposed study is to enhance the investigators understanding of the comprehensive psychosocial and medical needs of rural cancer patients and survivors along the cancer continuum, ultimately allowing us to address these gaps by identifying areas of support that can be bolstered by a population health navigator focused on rural populations.

DETAILED DESCRIPTION:
Primary objectives

To enhance understanding of the comprehensive psychosocial and medical needs of cancer survivors and caregivers in rural northwest North Carolina, focusing on their health needs, psychosocial concerns, perceived needs related to cancer and survivorship care, access/barriers to care, and knowledge/perceptions of clinical research using focus groups and semi-structured interviews. This aim is hypothesis-generating.

To document rural cancer patient/survivors' reports of: a) health behaviors; b) psychosocial needs; c) current health-related information and supportive care needs; d) barriers to care; e) symptoms and health-related quality of life using a quantitative survey

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis (other than non-melanoma skin cancer) and > 6 months post-definitive treatment (e.g., surgery, chemotherapy, and/or radiation); Survivors on ongoing systemic maintenance therapies (e.g., hormonal therapies and immunotherapies) are eligible
* Currently residing in one of the 6 priority counties in northwest North Carolina (Alleghany, Ashe, Avery, Mitchell, Stokes, Surry, Watauga, or Wilkes) or in a rural area in North Carolina as defined by a rural-urban commuting area (RUCA) code of 4-10.
* Ability and willingness to attend a one-time focus group or interview and/or complete a one-time study survey
* Age greater than 18 years.

Providers:

* Healthcare provider (e.g. primary care, oncology or other specialty, allied health) with knowledge of the needs of adult cancer survivors who are currently working in one of the priority counties in Northwest North Carolina (Alleghany, Ashe, Avery, Mitchell, Stokes, Surry, Watauga, or Wilkes)
* Ability and willingness to attend a one-time interview

Exclusion Criteria:

* Those who are unable to read and understand English, as the study interviews/focus groups and survey will be conducted in English
* Unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is adult men and women of all races and ethnicities who have received a diagnosis of cancer and are residing in a rural area of Northwest North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Improving Cancer-Related Experiences Through Interviews or Focus Group Settings | 90 minutes
  Through focus groups or interviews information will be collected on participants' experience receiving cancer-related care and to ask for specific suggestions and ways to improve care and cancer-related resources for adults living in a rural area.
Measurement of Quality of Life | 90 minutes
  The PROMIS Global 10 survey will be used to document rural cancer patient/survivors' reports of: a) health behaviors; b) psychosocial needs; c) current health-related information and supportive care needs; d) barriers to care; e) symptoms and health-related quality of life using a quantitative survey. Survey scoring consists of 5=Never, 4=Rarely, 3=Sometimes, 2=Often and 1=Always.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, MPH, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No